CLINICAL TRIAL: NCT06762769
Title: Isatuximab and Iberdomide as Immunotherapy for High Risk in Smouldering Myeloma
Acronym: MODIFY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Sanofi (Industry); Bristol Myers Squibb Pharmaceuticals Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/153707
Record Dates: First submitted 2024-12-09; First posted 2025-01-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-12

CONDITIONS: Smouldering Myeloma
Keywords: Isatuximab; Iberdomide; OBDS; Dexamethasone; MODIFY; Smouldering Myeloma; On Body Delivery System
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — isatuximab; iberdomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): All patients will receive 2 years of treatment, over 26 cycles. A cycle is 28 days. The treatment is split into 3 stages.
  Induction therapy: Cycle 1-4
  * Isatuximab is given once a week in cycle 1. Then twice a week in cycle 2-4. It is given subcutaneously using a medical device called an On Body Delivery System
  * Iberdomide is given on days 1-21. It is given as an oral capsule.
  * Dexamethasone is given once a week. It is given as an oral tablet.
  Consolidation therapy: Cycle 5-13
  * Isatuximab is given twice a week.
  * Iberdomide is given on days 1-21
  Maintenance therapy: Cycle 14-26
  * Isatuximab is given once a month
  * Iberdomide is given on days 1-21
  Interventions: Drug: Isatuximab; Drug: Iberdomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Subcutaneous isatuximab will be delivered using an unlicensed medical device (On Body Delivery System)
Drug: Iberdomide — Oral iberdomide
Drug: Dexamethasone — Oral dexamethasone

SUMMARY:
The study will test a new combination of 3 drugs: Isatuximab (Isa), Iberdomide (Iber) and Dexamethasone (Dex), in patients who have intermediate or high risk smouldering myeloma. Smouldering myeloma is an early form of myeloma which may progress to active multiple myeloma, but at a slow rate. Patients with smouldering myeloma do not usually receive any treatment but will have regular check-ups and observation. Some patients have a diagnosis of smouldering myeloma which has a higher risk of progressing to active myeloma.

The study will test if the combination of drugs is effective at preventing or delaying the disease progressing into active multiple myeloma. The study will also test if the combination is tolerated and accepted by patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and comply with protocol-mandated visits, treatment plan, laboratory tests and other study procedures.
2. Age ≥ 18 years
3. Diagnosed with smouldering myeloma (SMM) within 5 years of study registration AND diagnosed with intermediate or high risk SMM within 2 years of registration.:

   * i.e. patients may have been diagnosed de novo with intermediate or high risk smouldering myeloma within 2 years of study registration OR
   * patients may have been diagnosed with low or low-intermediate smouldering myeloma within 5 years of study registration and then their risk classification has changed to intermediate or high risk within 2 years of study registration.
4. Diagnosed with intermediate or high-risk SMM defined by IMWG diagnostic criteria and IMWG SMM risk stratification. Intermediate or high risk is defined by the presence of 2 or more of the following factors:

   * BM plasma cell infiltrate >20%
   * Serum paraprotein >20g/l
   * Serum Free Light Chain (SFLC) Ratio >20 (but <100)
   * Presence of t(4;14), t(14;16), del 17p, del 13q or 1q gain by fluorescence in situ hybridization (FISH) studies. Copy number abnormalities will be considered significant if present in ≥ 20% of cells.
5. Measurable disease with at least one of the following:

   * Paraprotein ≥5g/L
   * Serum free light chains ≥100mg/L with abnormal light chain ratio
   * Bence Jones protein ≥200mg/24hr
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
8. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 3 x ULN (if ALT and AST are tested, both must meet this criteria)
9. Adequate marrow function:

   * Neutrophils ≥1.0 x109/L (unless the participant has a known/suspected diagnosis of familial or racial neutropenia in which case an ANC ≥0.75 x 109/L is allowed),
   * Haemoglobin (Hb) ≥ 100g/L
   * Platelets ≥ 75 ×109/L
10. Creatinine clearance (CrCl) ≥ 30 mL/minute, according to the Cockcroft-Gault formula, following correction of reversible causes (e.g. dehydration, hypercalcaemia, sepsis)
11. Willing to comply with the contraceptive requirements of the trial

Exclusion Criteria:

1. Multiple Myeloma requiring treatment, as defined by IMWG SLiM-CRAB or CRAB criteria.
2. Monoclonal gammopathy of undetermined significance (MGUS), solitary plasmacytoma, primary amyloid light-chain (AL) amyloidosis.
3. Low or Low-intermediate risk smouldering myeloma by IMWG criteria
4. Received previous treatment for myeloma, smouldering myeloma or solitary plasmacytoma.
5. Treatment with any other standard anti-cancer radiotherapy/chemotherapy/targeted therapy including investigational therapy (defined as treatment for which there is currently no regulatory authority approved indication) within 4 weeks prior to registration.
6. Rapidly rising paraprotein or serum free light chains, defined as any of the following occurring within the space of 2 months:

   * doubling of serum M-protein (minimum rise 5g/l)
   * increase of serum M-protein by ≥10 g/L
   * increase of involved serum-free light chains (FLC) level by ≥200 mg/L (plus abnormal ratio)
   * increase of Bence Jones protein by ≥500mg/24hr
7. Corticosteroid treatment with a dose >10 mg prednisone or equivalent per day within 28 days of initiation of study drugs.
8. Unstable angina or myocardial infarction within 4 months prior to registration, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless patient has a pacemaker.
9. Prior or concurrent invasive malignancies except the following:

   * Adequately treated basal cell or squamous cell skin cancer.
   * Incidental finding of low grade (Gleason 3+3 or less) prostate cancer requiring no intervention. (Hormone monotherapy is permitted if overall survival is anticipated to be >5 years).
   * Adequately treated carcinoma in situ of the breast or cervix no longer requiring medical or surgical intervention.
   * Any cancer from which the patient has been disease-free for at least 3 years.
10. Any major surgery within 21 days prior to registration which in the investigator's opinion would compromise trial treatment and/or the patient's ability to comply with trial visits.
11. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of trial treatment, including difficulty swallowing.
12. Active systemic infection
13. Positive serologic and/or polymerase chain reaction (PCR) test results for acute or chronic hepatitis B virus (HBV) infection. (Note: Patients whose HBV infection status cannot be determined by serologic test results [see CDC website https://www.cdc.gov/hepatitis/hbv/pdfs/serologicchartv8.pdf] must be negative for HBV by PCR to be eligible for study participation). Patients with occult or prior HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable if they are willing to undergo DNA testing on Day 1 of every cycle and every three months for at least 12 months after the last cycle of study treatment and receive appropriate antiviral therapy.
14. Positive test results for hepatitis C virus (HCV). Note: Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation.
15. Positive test results for human immunodeficiency virus (HIV). Note: Patients with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy, have a CD4 count ≥ 200/μL, and have an undetectable viral load. HIV positive patients should be monitored per local/institutional standards while receiving study treatment.
16. Any other medical or psychiatric condition which, in the opinion of the investigator, contraindicates the participant's participation in this study.
17. Receipt of live vaccination within 30 days prior to registration, for the duration of the study and for 3 months after the last dose of study drug.
18. Contraindication to thromboprophylaxis.
19. Participant has risk factors for seizures or seizures that are not well controlled on current medication.
20. Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Treatment deliverability, measured by treatment discontinuation before completion of 26 cycles | From the date of registration until the date of treatment completion/discontinuation (approximately 2 years or earlier if patients discontinue treatment early)
  The number and proportion of patients who complete all 26 cycles of trial treatment per protocol (allowing for delays/reductions/omissions deemed acceptable by the protocol) will be presented with two-sided 90% confidence interval. While the sample size is based off of 57 patients being assessable for this endpoint, all eligible patients will be included in the analysis and conclusions will be based on the lower bound of the 90% confidence interval. Patients who do not complete treatment for reasons unrelated to disease or toxicity will be excluded from this analysis (e.g. patient moving away or becoming pregnant), however sensitivity analyses will be performed where these patients are assumed to complete/not complete treatment.
Treatment efficacy measured by best overall response rate by the end of treatment | From the date of registration until the date of 1 month follow up assessment
  The number and proportion of patients who achieve disease response (PR, VGPR, CR or sCR) at any point over the duration of treatment or at the 1 month FU response assessment will be presented with two-sided 90% confidence interval. While the sample size is based off of 53 patients being assessable for this endpoint, all eligible patients will be included in the analysis and conclusions will be based on the lower bound of the 90% confidence interval. All patients who have completed at least one response assessment or stopped protocol treatment early due to toxicity, insufficient response, progression or death will be included in this analysis.

SECONDARY OUTCOMES:
Progression Free Survival | From the date of registration until the date of first disease progression or death, whichever comes first, assessed up to 5.5 years
  PFS will be assessed using Kaplan-Meier survival analysis and will be defined as the time from registration until development of CRAB or SLiM CRAB or death from any cause. Patients who do not die or progress will be censored at the date of last adequate assessment with evidence of no progression (this will be at a minimum of 24 months for all patients who do not progress).
Time to biochemical progression | from the date of registration until the date of biochemical disease progression, assessed up to 5.5 years
  Time to biochemical progression will be assessed using Kaplan-Meier survival analysis and will defined as the time from registration until biochemical disease progression. Patients who do not have biochemical disease progression will be censored at the date last seen.
Progression Free Survival 2 | from the date of registration assessed up to 5.5 years
  PFS2 will be assessed using Kaplan-Meier survival analysis and will be measured in two ways:
  * from the date of registration until date of progression after diagnosis of active myeloma or death from any cause
  * from the date of progression to active myeloma to date of progression after diagnosis of active myeloma or death from any cause Patients who do not progress following diagnosis of active myeloma will be censored at the date last seen
Best overall response to subsequent line of therapy | From the date of registration until the end of follow up, assessed up to 5.5 years
  The best overall response rate to subsequent line of therapy will be presented with corresponding 95% confidence interval. Patients who do not start a new line of therapy will not be included in this analysis.
Overall Survival | From the date of registration until the date of death, assessed up to 5.5 years
  OS will be assessed using Kaplan-Meier survival analysis and will be defined as the time from registration until death from any cause. Patients who do not die will be censored at the date last seen
MRD negativity rates | From the date of screening until the date of 3 Years Post-Registration Follow Up
Very Good Partial Response and Complete response + MRD negative rates | From the date of screening until the date of 3 Years Post-Registration Follow Up
  Response rates (including PR, VGPR, CR, MRD negativity and VGPR/CR+MRD negativity) at each response assessment as well as best response over all assessments will be presented as the number and proportion with corresponding 95% confidence intervals. Patients who stopped treatment before the response assessment due to toxicity, insufficient response, progression or death will be counted as non-responders.
Adverse Event and Adverse Device Effect rates | From informed consent until the end of post-treatment safety reporting window (6 months after the last dose)
  Assessed by CTCAE criteria v5. Assessed in all patients given at least one dose of study treatment.
  The worst grade of each adverse event and adverse device effect for each patient will be calculated and the rates of grade 1-2 and 3-5 will be summarised. Analyses looking at the number of each AE and ADE experienced by patients and the duration of symptoms will also be considered to assess the entire burden of toxicity. Toxicity data Separate analyses will be summarised across the entire duration of treatment as well as by treatment phase performed using a) all toxicity data and b) toxicity data during cycles 1-4 (induction, consolidation, maintenance) only.).
Median and cumulative doses of Iberdomide and Isatuximab | From registration until end of treatment (approximately 2 years or earlier if patients discontinue treatment early)
Treatment compliance | From registration until end of treatment (approximately 2 years or earlier if patients discontinue treatment early)
  The treatment discontinuation rates during each phase of treatment (Induction cycles 1-4; Consolidation cycles 5-13 and Maintenance cycles 14-26) will be presented with corresponding 95% confidence intervals.
Patient Reported Outcome Measures (EORTC QLQ-C30) | From the date of screening until the date of progression or Month 12 Follow up visit, whichever is latest
  Quality of life data will be summarised using descriptive statistics and plotted over time to describe any changes throughout treatment and follow up
Patient Reported Outcome Measures (EORTC QLQ-MY20) | From the date of screening until the date of progression or Month 12 Follow up visit, whichever is latest
  Quality of life data will be summarised using descriptive statistics and plotted over time to describe any changes throughout treatment and follow up.
Patient Reported Outcome Measures (EQ5D-3L) | From the date of screening until the date of progression or Month 12 Follow up visit, whichever is latest
  Quality of life data will be summarised using descriptive statistics and plotted over time to describe any changes throughout treatment and follow up
Patient Reported Outcome Measures (Bespoke MODIFY questionnaire) | From the date of screening until the date of progression or Month 12 Follow up visit, whichever is latest
  Quality of life data will be summarised using descriptive statistics and plotted over time to describe any changes throughout treatment and follow up

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Barts Health Trust, London
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No